CLINICAL TRIAL: NCT00567723
Title: A Phase-IV, Long-term, Observational Safety Study in End Stage Renal Disease Subjects Treated With Lanthanum Carbonate (Fosrenol)
Brief Title: Long Term Treatment of End Stage Renal Disease Patients With Lanthanum Carbonate (Fosrenol)
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SPD405-404
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Test group: Patients who have received a minimum of 12 consecutive weeks of treatment with Fosrenol
- 2: Historical control group: Patients with no lanthanum exposure
- 3: Concomitant therapy group: Patients being treated for hyperphosphatemia with any marketed product

SUMMARY:
Patients who have been treated with Fosrenol for a minimum of 12 consecutive weeks and are receiving dialysis will be followed for 5 years to compare mortality, bone fractures and incidence of selected morbidities to patients with no lanthanum exposure and to patients being treated for hyperphosphatemia with any marketed product.

ELIGIBILITY:
Inclusion Criteria: Test Group

* Signed informed consent
* Patient must have ESRD and be receiving dialysis
* Prior treatment with Fosrenol for a minimum of 12 consecutive weeks
* Primary payer of healthcare must be Medicare (patient must supply Medicare Claim Number)
* Patient must be 18 years of age or older

Exclusion Criteria: Test Group

* Patients that do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for the Historical Control and Concomitant Therapy Groups will be selected from the United States Renal Data System (USRDS). The Test Group will consist of patients who have had a minimum of 12 consecutive weeks of exposure to Fosrenol (lanthanum carbonate).
Sampling Method: Probability Sample
Enrollment: 2105 (Actual)
Dates: Start 2006-04-25 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-07 (Actual)

PRIMARY OUTCOMES:
Compare all-cause mortality and bone fractures among three groups of subjects with end stage renal disease (ESRD) | 5 years

SECONDARY OUTCOMES:
Compare the incidence of selected morbidities among three groups of patients with ESRD | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (195):
- United States (195):
  - Clinical Research Center, Inc., Birmingham, Alabama
  - Clinical Research Consultants, Hoover, Alabama
  - University of South Alabama, Mobile, Alabama
  - Montgomery Kidney Specialists, Montgomery, Alabama
  - California Kidney Specialist, Covina, California
  - Atlantic Avenue Medical Clinic, Cudahy, California
  - East Bay-South Hayward Dialysis Center, Hayward, California
  - Renal Research Center, Los Alamitos, California
  - USC Kidney Center, Los Angeles, California
  - Beverly Nephrology, Los Angeles, California
  - Tower Nephrology Medical Group, Los Angeles, California
  - USC DaVita Dialysis Center, Los Angeles, California
  - Renal Medical Associates, Lynwood, California
  - Valley Renal Medical Group, Northridge, California
  - Desert Nephrolgy Medical Group, Palm Springs, California
  - Palo Alto Nephrology, Palo Alto, California
  - Pasadena Nephrology, Pasadena, California
  - Capital Nephrology, Sacramento, California
  - Citrus Valley Dialysis Center, San Bernardino, California
  - California Kidney Specialist, San Dimas, California
  - San Francisco Dialysis Center # 3830, San Francisco, California
  - Habib A. Tobbagi, MD, San Jose, California
  - Selma DaVita Dialysis, Selma, California
  - Pear Tree Dialysis, Ukiah, California
  - High Desert Nephrology, Victorville, California
  - Renal Medical Group, Visalia, California
  - North Valley Nephrology, Yuba City, California
  - Hartford North, Hartford, Connecticut
  - Metabolism Associates, New Haven, Connecticut
  - Torrington Dialysis, Torrington, Connecticut
  - Davita-Brentwood, Washington D.C., District of Columbia
  - Lee Street Dialysis, Washington D.C., District of Columbia
  - Union Plaza Dialysis Center, Washington D.C., District of Columbia
  - PAB Clinical Resesarch, Brandon, Florida
  - South Florida Nephrology Group, Coral Springs, Florida
  - Nephrology Consultants, PA, Daytona Beach, Florida
  - DaVita Fort Myers, Fort Myers, Florida
  - Nephrology Associates, Ft. Pierce, Florida
  - Outcomes Research International, Inc, Hudson, Florida
  - Central Florida Kidney Care, PA, Lakeland, Florida
  - Miami Kidney Group, Miami, Florida
  - Nephrology Associates of South Miami, Miami, Florida
  - Nephrology Associates of Central Florida, Orlando, Florida
  - Nephrology Associates Research Center, Panama City, Florida
  - A Unique Kidney Center, LLC, Pembroke Pines, Florida
  - PharmResearch, Inc., Pinecrest, Florida
  - Tampa Bay Nephrology Associates, Tampa, Florida
  - Genesis Clinical Research, Tampa, Florida
  - North Georgia Nephrology Consultant, Athens, Georgia
  - Southwest Atlanta Nephrology, PC, Atlanta, Georgia
  - North Atlantic Kidney Specialist, Atlanta, Georgia
  - AtlantaDavita East, Atlanta, Georgia
  - Davita South Fulton, Atlanta, Georgia
  - Kidney Care Associates, LLC, Augusta, Georgia
  - Douglas Dialysis, Douglas, Georgia
  - Renal Physicians of Georgia, Dublin, Georgia
  - Renal Physicians of Georgia, Macon, Georgia
  - Williams Street Dialysis, Savannah, Georgia
  - Waycross Dialysis Facility, Waycross, Georgia
  - Table Rock Dialysis, Boise, Idaho
  - Nampa DaVita Dialysis, Nampa, Idaho
  - Fox Valley Dialysis, Aurora, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Associates in Nephrology, Des Plaines, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Associates in Nephrology, Evergreen Park, Illinois
  - North Suburban Nephrology, LLC, Gurnee, Illinois
  - Lake County, Libertyville, Illinois
  - Nephrology & Hypertension Consultants, PC, Park Ridge, Illinois
  - Renal Care Associates, Peoria, Illinois
  - Sauget Dialysis, Sauget, Illinois
  - Nephrology Associates, LLC, Evansville, Indiana
  - Nephrology Specialists PC, Gary, Indiana
  - Lawrenceburg Dialysis Center, Lawrenceburg, Indiana
  - Nephrology Specialists, Michigan City, Indiana
  - Renal Associates of Central Indiana, Muncie, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - TriMark Physicians Group, Fort Dodge, Iowa
  - Olathe DaVita, Olathe, Kansas
  - DaVita-Johnson County Dialysis, Overland Park, Kansas
  - Veritas Clinical Specialists, Ltd, Topeka, Kansas
  - Dennis Artzer, Topeka, Kansas
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - West Bank Nephrology, Marrero, Louisiana
  - LSU Healthcare Network, New Orleans, Louisiana
  - Westbank Chronic Renal Center, New Orleans, Louisiana
  - Northwest Louisiana Nephrology, LLC, Shreveport, Louisiana
  - DaVita JHHS Bond Street, Baltimore, Maryland
  - Nephrology and Hypertension, Clinton, Maryland
  - DaVita Frederick Dialysis #3373, Frederick, Maryland
  - Glen Burnie Dialysis Center, Glen Burnie, Maryland
  - Promod K. Duggal, MD, PC, Greenbelt, Maryland
  - Rivertowne Davita Dialysis, Oxon Hill, Maryland
  - Biolab Research, LLC, Rockville, Maryland
  - Davita of Landover, Upper Marlboro, Maryland
  - Carroll County Dialysis Facility, Westminster, Maryland
  - Horowitz and Krahn, Fall River, Massachusetts
  - Western New England Renal Transplant Association, Springfield, Massachusetts
  - Great Lakes Renal Network, Alma, Michigan
  - PDI Grand Rapids East, Grand Rapids, Michigan
  - Mid Michigan Kidney Specialists, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Macomb Kidney Center, Warren, Michigan
  - Health Sciences Center, Columbia, Missouri
  - Douglas T. Domoto MD, JD, PC, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Louis University Department of Internal Medicine, St Louis, Missouri
  - Hypertension & Nephrology Associates, PA, Eatontown, New Jersey
  - DaVita Edison, Edison, New Jersey
  - Center for Kidney Care, Mount Laurel, New Jersey
  - Cumberland Nephrology Associates, PA, Vineland, New Jersey
  - Kidney Care Associates, PLLC, Brooklyn, New York
  - Angelo Magno, MD, Brooklyn, New York
  - Brookdale Physicians Dialysis associates, P.C., Brooklyn, New York
  - Celia Dill Dialysis Center, Carmel, New York
  - AMS Research, Elmira, New York
  - Nephrology Associates, PC, Flushing, New York
  - North Shore University Hospital, Great Neck, New York
  - Lower Manhattan Dialysis Center, New York, New York
  - Bronx Dialysis center, New York, New York
  - Nephrology Associates, Rochester, New York
  - University of Rochester Nephrology Unit, Rochester, New York
  - Island Renal Associates, PC, Rockville Centre, New York
  - Clinical Research Development Association, LLC, Springfield Gardens, New York
  - SUNY at Stony Brook NY, Stony Brook, New York
  - Syosset Kidney Center, Syosset, New York
  - Yonkers Nephrology, PC, Yonkers, New York
  - Mountain Kidney, Asheville, North Carolina
  - University of North Carolina Division of Nephrology & Hypertension, Chapel Hill, North Carolina
  - Charlotte Dialysis, Charlotte, North Carolina
  - Albemarle Nephrology Associates, Elizabeth City, North Carolina
  - Dialysis Care of Richmond County, Hamlet, North Carolina
  - Dialysis Care of Hoke County, Raeford, North Carolina
  - Reidsville Dialysis, Reidsville, North Carolina
  - Southeastern Nephrology Associates, Wilmington, North Carolina
  - DaVita Wilson Dialysis #3032, Wilson, North Carolina
  - Nephrology Associates, PLLC, Winston-Salem, North Carolina
  - Altru Health System Research Center, Grand Forks, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Nephrology Consultants of Northwest Ohio, Toledo, Ohio
  - Saint Elizabeth Healthcare Department of Research, Youngstown, Ohio
  - NAI fo Kidney Care, Youngstown, Ohio
  - Nephrology Assciates of Central PA, INC, Camp Hill, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Renal Care of Erie, Erie, Pennsylvania
  - Exton Dialysis Center, Exton, Pennsylvania
  - Davita Lancaster, Lancaster, Pennsylvania
  - Lewistown Dialysis Center, Lewistown, Pennsylvania
  - Reading Nephrology, Ltd., Mohnton, Pennsylvania
  - Pennyslvania Nephrology Associates, PC, Philadelphia, Pennsylvania
  - Davita West Philadelphia, Philadelphia, Pennsylvania
  - Franklin Dialysis Center, Philadelphia, Pennsylvania
  - Syed Shah, Pottsville, Pennsylvania
  - Syed Shah, Saint Clair, Pennsylvania
  - Washington Dialysis, Washington, Pennsylvania
  - Dialyis Corporation of America, Wellsboro, Pennsylvania
  - Reading Nephrology, Ltd., West Reading, Pennsylvania
  - Reading Nephrology, Ltd, Wyomissing, Pennsylvania
  - Nephrology and Internal Medicine, Anderson, South Carolina
  - Carolina Nephrology, PA, Greenville, South Carolina
  - Internal Medicine Nephrology/Hypertension, Kingstree, South Carolina
  - Charleston Nephrology Associates, North Charleston, South Carolina
  - Southern Pines Dialysis, Southern Pines, South Carolina
  - Newman, Knoxville, Tennessee
  - G. Edward Newman, MD, PLLC, Knoxville, Tennessee
  - Internal Medicina and Nephrology, Maynardville, Tennessee
  - Memphis Central DaVita, Memphis, Tennessee
  - VA Tennessee Valley, Health Care System, Nashville, Tennessee
  - Arlington Nephrology, PA, Arlington, Texas
  - Brenham, Brenham, Texas
  - Kidney Consultants fo El Paso, P.A., El Paso, Texas
  - Med-Center Dialysis, Houston, Texas
  - Innovative Renal Care, Houston, Texas
  - Northwest Kidney Center, Houston, Texas
  - Greater Houston Kidney Specialist, Houston, Texas
  - Kidney Associates, PLLC, Houston, Texas
  - DaVita Northstar Dialysis, Houston, Texas
  - Patel, Wichita Falls, Texas
  - Pharmaceutical Research Organization, Bountiful, Utah
  - Nephrology of Northern Utah, Ogden, Utah
  - Central Utah Clinic, Provo, Utah
  - University of Vermont, Fletcher Allen Health Care, Burlington, Vermont
  - Jefferson Nephrology Ltd, Charlottesville, Virginia
  - Great Bridge Dialysis Center, Chesapeake, Virginia
  - Nephrology Associates of Northern Virgina, Fairfax, Virginia
  - Piedmont Medical and Renal Associates, Martinsville, Virginia
  - Peninsula Dialysis, Newport News, Virginia
  - Davita-Greater Portsmouth, Portsmouth, Virginia
  - Portsmouth Dialysis Center-DaVita, Portsmouth, Virginia
  - Nephrology Specialists, PC, Richmond, Virginia
  - Lakewood Community Dialysis Center, Lakewood, Washington
  - Fox Valley Nephrology Partners, SC, Appleton, Wisconsin
  - Purity Dialysis Centers, Delafield, Wisconsin
  - Gundersen Lutheran, Ltd, La Crosse, Wisconsin
  - Fox Valley Nephrology Partners, PC, Oshkosh, Wisconsin

REFERENCES:
- [Derived] Hutchison A, Whelton A, Thadhani R, Achenbach H, Vergani A, Wu J, Hall G. Long-Term Mortality and Bone Safety in Patients with End-Stage Renal Disease Receiving Lanthanum Carbonate. Nephron. 2018;140(4):265-274. doi: 10.1159/000492603. Epub 2018 Oct 23. PMID 30352437
- [Derived] Hutchison AJ, Wilson RJ, Garafola S, Copley JB. Lanthanum carbonate: safety data after 10 years. Nephrology (Carlton). 2016 Dec;21(12):987-994. doi: 10.1111/nep.12864. PMID 27479781
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5feb4db2bf003ab47c4a